CLINICAL TRIAL: NCT02817672
Title: Scaling a Smarter and More Efficient Intervention: Evaluating the Feasibility of Disseminating a Novel Mobile App Platform to Treat Depression
Brief Title: Evaluating the Feasibility of Disseminating a Novel Mobile Platform to Treat Depression
Acronym: PRIME-D
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The dataset was not strong enough to do NLP analysis.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH110583-01 (NIH)
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Depression
Keywords: Human; Mental Disorders; intervention; digital health
MeSH Terms: conditions — Depression; Mental Disorders | interventions — prime and bond 2.0

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- PRIME 1.0 (Active Comparator): 8 weeks use of PRIME 1.0 (current version). Mobile application designed to improve psychosocial functioning and motivational deficits.
  Interventions: Behavioral: PRIME 1.0
- PRIME 2.0 (Experimental): 8 weeks use of PRIME 2.0 (version with the NLP-powered dashboard). Mobile application designed to improve psychosocial functioning and motivational deficits.
  Interventions: Behavioral: PRIME 2.0

INTERVENTIONS:
Behavioral: PRIME 1.0 — Mobile application designed to improve psychosocial functioning and motivational deficits (sans NLP-powered dashboard).
  Arms: PRIME 1.0
Behavioral: PRIME 2.0 — Mobile application designed to improve psychosocial functioning and motivational deficits (with NLP-powered dashboard).
  Arms: PRIME 2.0

SUMMARY:
The goal of this project is to conduct a pilot study to test the utility of a Natural Language Processing (NLP) clinical messaging tool to improve the reach and the quality (fidelity and competency) of coaches providing behavioral activation (BA) strategies through a mobile mental health app called Personalized Real-time Intervention for Motivational Enhancement (PRIME). This study will improve the reach of clinicians by using a NLP-powered messaging tool, which will ensure fidelity to the BA model and clinicians will have access to real-time clinical information about their patients to guide more targeted treatment (competence). If successful, PRIME could operate as a cost effective tool for clinicians to extend their reach and an accessible treatment for the population of those struggling with depression.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Read and speak English
* PHQ-9 score of 5 or greater or indicate that their depressive symptoms are interfering with their daily functioning (Item 10 of the PHQ-9 > 2).
* To be consistent with the NIMH RDoC initiative, we will assess for co-morbid problems (substance abuse, anxiety, and psychosis), but will not exclude participants with psychiatric comorbidities
* Must own a mobile device on iOS or Android platforms that either Wi-Fi or 3G/4G ready;

Exclusion Criteria:

* Under 18
* Cannot read or speak in English
* Cannot attain suitable mobile device

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Depression severity | Change from baseline to 3 month follow-up
  PhQ-9
Functioning | Change from baseline to 3 month follow-up
  Sheehan Disability Scale

SECONDARY OUTCOMES:
Coaching efficiency | 8 weeks
  Flurry analytics
Coaching competence | 8 weeks
  Fidelity and competence assessment

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Schlosser, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Schlosser D, Campellone T, Kim D, Truong B, Vergani S, Ward C, Vinogradov S. Feasibility of PRIME: A Cognitive Neuroscience-Informed Mobile App Intervention to Enhance Motivated Behavior and Improve Quality of Life in Recent Onset Schizophrenia. JMIR Res Protoc. 2016 Apr 28;5(2):e77. doi: 10.2196/resprot.5450. PMID 27125771
- [Background] Fisher M, Loewy R, Hardy K, Schlosser D, Vinogradov S. Cognitive interventions targeting brain plasticity in the prodromal and early phases of schizophrenia. Annu Rev Clin Psychol. 2013;9:435-63. doi: 10.1146/annurev-clinpsy-032511-143134. Epub 2013 Jan 7. PMID 23297786